CLINICAL TRIAL: NCT06466733
Title: Puerto Rico Embolization of the Middle Meningeal Artery for the Treatment of Chronic Subdural Hematoma Trial (PREMMA)
Acronym: PREMMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan M. Ramos Acevedo (Other)
Responsible Party: Sponsor-Investigator, Juan M. Ramos Acevedo, Principal Investigator, University of Puerto Rico
Organization: University of Puerto Rico (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2305109135
Record Dates: First submitted 2024-05-15; First posted 2024-06-20 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Embolization of the middle meningeal artery; Surgical evacuation; Hemorrhage; Intracranial hemorrhage; Cerebrovascular disease; Chronic disease
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hemorrhage; Intracranial Hemorrhages; Cerebrovascular Disorders; Chronic Disease | interventions — Craniotomy; Trephining

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endovascular Embolization (Experimental): Embolization of the middle meningeal artery
  Interventions: Procedure: Embolization of the middle meningeal artery
- Surgical Evacuation of Hematoma (Active Comparator): Burr hole or craniotomy
  Interventions: Procedure: Surgical Evacuation via burr hole or craniotomy

INTERVENTIONS:
Procedure: Embolization of the middle meningeal artery — Embolization of the middle meningeal artery ipsilateral to the chronic subdural hematoma is performed infusing embolic polyvinyl alcohol (PVA) microparticles.
  Arms: Endovascular Embolization
Procedure: Surgical Evacuation via burr hole or craniotomy — The standard of care for chronic subdural hematoma, burr hole or craniotomy are performed ipsilateral to the lesion.
  Other Names: Burr hole; Craniotomy
  Arms: Surgical Evacuation of Hematoma

SUMMARY:
Puerto Rico Embolization of the Middle Meningeal Artery (PREMMA) trial is a multi-center, parallel, prospective, superiority, randomized controlled trial with concealed allocation comparing reoperation rates and neurological outcomes in patients with chronic subdural hematoma that receive treatment via embolization of the middle meningeal artery versus surgical evacuation via burr hole trephination or craniotomy.

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is a collection of fluid and blood breakdown products that evolves over weeks to months in the subdural space. This condition is more common among people older than 65 years and has been associated with increased use of antithrombotic therapy among this population. The World population is rapidly aging; thus, the investigators expect the number of patients with cSDH will increase. The United Nations World Social Report places Puerto Rico in the 7th place of countries with the largest share of people aged 65 years or over. This pathology burdens healthcare systems; therefore, assessing the feasibility of treatment modalities for cSDH that are less invasive, have lower procedural risks, and have lower recurrence rates that require additional surgical intervention is essential.

The standard of care for symptomatic cSDH is the surgical evacuation (SE) of the hematoma, with recurrence rates between 10-30% and surgical rescue indicated for most of these cases. Evacuation of the hematoma effectively relieves its mass effect but does not change the underlying pathophysiologic mechanism. In recent years, embolization of the middle meningeal artery (eMMA) has been shown to decrease the recurrence of chronic subdural hematoma and the need for revision burr hole or craniotomy. The PREMMA trial aims to compare embolization of the middle meningeal artery as stand-alone treatment for chronic subdural hematoma versus the standard of care, surgical evacuation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Speak and understand Spanish or English
* Resident of Puerto Rico
* Glasgow coma scale ≥ 14/15
* Presence of cSDH on non-contrast computed tomography (NCCT) or magnetic resonance imaging (MRI)
* Neurological indication for treatment of cSDH (Markwalder scale ≤ 2)
* No previous surgical or endovascular treatment for symptomatic cSDH
* Signed informed consent for participation in the study by the patient or legally authorized representative

Exclusion Criteria:

* Acute subdural hematoma
* Focal, non-hemispheric localization of cSDH
* Evidence of other lesions associated with cSDH, such as neoplasms, vascular lesions, or additional epidural, subarachnoid, or parenchymal hemorrhage on non-contrast computed tomography or magnetic resonance imaging
* Imaging evidence of skull fracture over the subdural hematoma
* Presence of any cerebrospinal fluid (CSF) shunt
* Imaging evidence of midline shift ≥ 10 mm
* Imaging evidence of basal cistern effacement
* Imaging evidence of dilatation of lateral ventricles
* Imaging evidence of uncal herniation
* Modified Rankin scale ≥ 3 before developing symptoms associated with cSDH
* Contraindications for angiography (i.e., complex anatomy or kidney failure)
* Comorbidity making follow-up impossible
* Pregnancy
* Vulnerable patients, including homeless patients, incarcerated patients, and mentally ill patients without appropriate medical decision-making proxies that the physician believes are incapable of appropriately assessing the risks of the procedure
* Absence of medical insurance

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Reoperation | 3 months, 6 months, and 12 months
  Number of patients requiring reoperation due to recurrent chronic subdural hematoma.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | Pre-operative, 24 hours, 2 weeks, 1.5 months, 3 months, 6 months, and 12 months
  The modified Rankin Scale (mRS) will assess neurological disability. The scale comprises seven levels, from 0 to 6, with higher scores indicating greater disability, and 6 indicating death.
Glasgow Coma Scale (GCS) | Pre-operative, 24 hours, 2 weeks
  The Glasgow coma scale (GCS) will assess consciousness level. GCS score can range from 3 (completely unresponsive) to 15 (completely alert and oriented).
Visual Analog Scale (VAS) | Pre-operative, 24 hours, 2 weeks, 1.5 months, 3 months, 6 months, 12 months
  The visual analog scale (VAS) will assess pain levels. VAS represents the severity of pain from 0 "no pain" to 10 "very severe pain."
Quality of life (EQ-5D-5L) | Pre-operative, 2 weeks, 1.5 months, 3 months, 6 months, 12 months
  Will be measured with the EuroQol 5 dimensions and 5 levels (EQ-5D-5L) grading scale.
Radiological outcomes | Pre-operative, 24 hours, 3 months, 6 months, 12 months
  Will be measured by routine computed tomography compared with pre-operative images.
Technical success of embolization of the middle meningeal artery (eMMA) | 24 hours
  The rate of unsuccessful eMMA due to technical failure or anatomical issues will be recorded.
Procedure-related complications | 24 hours, 2 weeks, 1.5 months, 3 months
  Any life-threatening event from enrollment to discharge will be recorded.
Adverse events | 24 hours, 2 weeks, 1.5 months, 3 months
  Any unintentional injury or complication involving a prolonged stay, disability at discharge, or death caused by healthcare management, not the underlying disease, will be recorded.
Post-operative morbidity | 24 hours, 2 weeks, 1.5 months, 3 months
  All surgical and/or medical complications that occur.
Mortality | 24 hours, 2 weeks, 30 days, 1.5 months, 3 months, 6 months, 12 months
  The number of participants among the total number of deaths.
Length of stay | From date of randomization until the date of discharge or date of death from any cause while patient is in hospital, whichever came first, assessed up to 90 days
  The patient's hospitalization period.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Ramos Acevedo, MD, Principal Investigator — University of Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ropper AH. Beneath a Tough Mother (Dura Mater) - Chronic Subdural Hematoma. N Engl J Med. 2020 Dec 31;383(27):2678-2680. doi: 10.1056/NEJMe2031257. Epub 2020 Dec 16. No abstract available. PMID 33326714
- [Background] Jung YG, Jung NY, Kim E. Independent predictors for recurrence of chronic subdural hematoma. J Korean Neurosurg Soc. 2015 Apr;57(4):266-70. doi: 10.3340/jkns.2015.57.4.266. Epub 2015 Apr 24. No abstract available. PMID 25932293
- [Background] Edlmann E, Giorgi-Coll S, Whitfield PC, Carpenter KLH, Hutchinson PJ. Pathophysiology of chronic subdural haematoma: inflammation, angiogenesis and implications for pharmacotherapy. J Neuroinflammation. 2017 May 30;14(1):108. doi: 10.1186/s12974-017-0881-y. PMID 28558815
- [Background] Moshayedi P, Liebeskind DS. Middle Meningeal Artery Embolization in Chronic Subdural Hematoma: Implications of Pathophysiology in Trial Design. Front Neurol. 2020 Aug 27;11:923. doi: 10.3389/fneur.2020.00923. eCollection 2020. PMID 32973670
- [Background] Henry J, Amoo M, Kissner M, Deane T, Zilani G, Crockett MT, Javadpour M. Management of Chronic Subdural Hematoma: A Systematic Review and Component Network Meta-analysis of 455 Studies With 103 645 Cases. Neurosurgery. 2022 Dec 1;91(6):842-855. doi: 10.1227/neu.0000000000002144. Epub 2022 Sep 28. PMID 36170165
- [Background] Dudoit T, Labeyrie PE, Deryckere S, Emery E, Gaberel T. Is systematic post-operative CT scan indicated after chronic subdural hematoma surgery? A case-control study. Acta Neurochir (Wien). 2016 Jul;158(7):1241-6. doi: 10.1007/s00701-016-2820-6. Epub 2016 May 5. PMID 27147520
- [Background] Chen FM, Wang K, Xu KL, Wang L, Zhan TX, Cheng F, Wang H, Chen ZB, Gao L, Yang XF. Predictors of acute intracranial hemorrhage and recurrence of chronic subdural hematoma following burr hole drainage. BMC Neurol. 2020 Mar 13;20(1):92. doi: 10.1186/s12883-020-01669-5. PMID 32169039
- [Background] Thomas PAW, Mitchell PS, Marshman LAG. Early Postoperative Morbidity After Chronic Subdural Hematoma: Predictive Usefulness of the Physiological and Operative Severity Score for Enumeration of Mortality and Morbidity, American College of Surgeons National Surgical Quality Improvement Program, and American Society of Anesthesiologists Grade in a Prospective Cohort. World Neurosurg. 2019 Apr;124:e489-e497. doi: 10.1016/j.wneu.2018.12.119. Epub 2019 Jan 3. PMID 30610985
- [Background] Kolias AG, Chari A, Santarius T, Hutchinson PJ. Chronic subdural haematoma: modern management and emerging therapies. Nat Rev Neurol. 2014 Oct;10(10):570-8. doi: 10.1038/nrneurol.2014.163. Epub 2014 Sep 16. PMID 25224156
- [Background] Santarius T, Kirkpatrick PJ, Ganesan D, Chia HL, Jalloh I, Smielewski P, Richards HK, Marcus H, Parker RA, Price SJ, Kirollos RW, Pickard JD, Hutchinson PJ. Use of drains versus no drains after burr-hole evacuation of chronic subdural haematoma: a randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1067-73. doi: 10.1016/S0140-6736(09)61115-6. PMID 19782872
- [Background] Nouri A, Gondar R, Schaller K, Meling T. Chronic Subdural Hematoma (cSDH): A review of the current state of the art. Brain Spine. 2021 Nov 2;1:100300. doi: 10.1016/j.bas.2021.100300. eCollection 2021. PMID 36247395
- [Background] Desir LL, Narayan V, Ellis J, Gordon D, Langer D, Ortiz R, Serulle Y. Middle Meningeal Artery Embolization in the Management of Chronic Subdural Hematoma: a Comprehensive Review of Current Literature. Curr Neurol Neurosci Rep. 2023 Apr;23(4):109-119. doi: 10.1007/s11910-023-01262-6. Epub 2023 Apr 11. PMID 37037979
- [Background] Miah IP, Tank Y, Rosendaal FR, Peul WC, Dammers R, Lingsma HF, den Hertog HM, Jellema K, van der Gaag NA; Dutch Chronic Subdural Hematoma Research Group. Radiological prognostic factors of chronic subdural hematoma recurrence: a systematic review and meta-analysis. Neuroradiology. 2021 Jan;63(1):27-40. doi: 10.1007/s00234-020-02558-x. Epub 2020 Oct 22. PMID 33094383
- [Background] Rauhala M, Helen P, Huhtala H, Heikkila P, Iverson GL, Niskakangas T, Ohman J, Luoto TM. Chronic subdural hematoma-incidence, complications, and financial impact. Acta Neurochir (Wien). 2020 Sep;162(9):2033-2043. doi: 10.1007/s00701-020-04398-3. Epub 2020 Jun 10. PMID 32524244
- [Background] Almenawer SA, Farrokhyar F, Hong C, Alhazzani W, Manoranjan B, Yarascavitch B, Arjmand P, Baronia B, Reddy K, Murty N, Singh S. Chronic subdural hematoma management: a systematic review and meta-analysis of 34,829 patients. Ann Surg. 2014 Mar;259(3):449-57. doi: 10.1097/SLA.0000000000000255. PMID 24096761
- [Background] Ironside N, Nguyen C, Do Q, Ugiliweneza B, Chen CJ, Sieg EP, James RF, Ding D. Middle meningeal artery embolization for chronic subdural hematoma: a systematic review and meta-analysis. J Neurointerv Surg. 2021 Oct;13(10):951-957. doi: 10.1136/neurintsurg-2021-017352. Epub 2021 Jun 30. PMID 34193592
- [Background] Mignucci-Jimenez G, Matos-Cruz AJ, Abramov I, Hanalioglu S, Kovacs MS, Preul MC, Feliciano-Valls CE. Puerto Rico Recurrence Scale: Predicting chronic subdural hematoma recurrence risk after initial surgical drainage. Surg Neurol Int. 2022 Jun 3;13:230. doi: 10.25259/SNI_240_2022. eCollection 2022. PMID 35855136
- [Background] Flores G, Vicenty JC, Pastrana EA. Post-operative seizures after burr hole evacuation of chronic subdural hematomas: is prophylactic anti-epileptic medication needed? Acta Neurochir (Wien). 2017 Nov;159(11):2033-2036. doi: 10.1007/s00701-017-3298-6. Epub 2017 Aug 15. PMID 28808801
- [Background] De Jesus O, Pacheco H, Negron B. Chronic and subacute subdural hematoma in the adult population. The Puerto Rico experience. P R Health Sci J. 1998 Sep;17(3):227-33. PMID 9883468
- [Background] De Jesus O, Monserrate AE. Burr Hole Surgery for Drainage of Chronic and Subacute Subdural Hematomas: Low Recurrence Rate in a Single Surgeon Cohort. Cureus. 2021 Nov 5;13(11):e19288. doi: 10.7759/cureus.19288. eCollection 2021 Nov. PMID 34900470
- [Background] Altaf I, Shams S, Vohra AH. Radiolological predictors of recurrence of chronic subdural hematoma. Pak J Med Sci. 2018 Jan-Feb;34(1):194-197. doi: 10.12669/pjms.341.13735. PMID 29643906
- [Background] Joyce E, Bounajem MT, Scoville J, Thomas AJ, Ogilvy CS, Riina HA, Tanweer O, Levy EI, Spiotta AM, Gross BA, Jankowitz BT, Cawley CM, Khalessi AA, Pandey AS, Ringer AJ, Hanel R, Ortiz RA, Langer D, Levitt MR, Binning M, Taussky P, Kan P, Grandhi R. Middle meningeal artery embolization treatment of nonacute subdural hematomas in the elderly: a multiinstitutional experience of 151 cases. Neurosurg Focus. 2020 Oct;49(4):E5. doi: 10.3171/2020.7.FOCUS20518. PMID 33002874
- [Background] Ban SP, Hwang G, Byoun HS, Kim T, Lee SU, Bang JS, Han JH, Kim CY, Kwon OK, Oh CW. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma. Radiology. 2018 Mar;286(3):992-999. doi: 10.1148/radiol.2017170053. Epub 2017 Oct 10. PMID 29019449
- [Background] Desir LL, D'Amico R, Link T, Silva D, Ellis JA, Doron O, Langer DJ, Ortiz R, Serulle Y. Middle Meningeal Artery Embolization and the Treatment of a Chronic Subdural Hematoma. Cureus. 2021 Oct 18;13(10):e18868. doi: 10.7759/cureus.18868. eCollection 2021 Oct. PMID 34754700
- [Background] Ashry A, Al-Shami H, Gamal M, Salah AM. Local anesthesia versus general anesthesia for evacuation of chronic subdural hematoma in elderly patients above 70 years old. Surg Neurol Int. 2022 Jan 12;13:13. doi: 10.25259/SNI_425_2021. eCollection 2022. PMID 35127213
- [Background] Catapano JS, Ducruet AF, Nguyen CL, Cole TS, Baranoski JF, Majmundar N, Wilkinson DA, Fredrickson VL, Cavalcanti DD, Lawton MT, Albuquerque FC. A propensity-adjusted comparison of middle meningeal artery embolization versus conventional therapy for chronic subdural hematomas. J Neurosurg. 2021 Feb 26;135(4):1208-1213. doi: 10.3171/2020.9.JNS202781. Print 2021 Oct 1. PMID 33636706
- [Background] Dian J, Linton J, Shankar JJ. Risk of recurrence of subdural hematoma after EMMA vs surgical drainage - Systematic review and meta-analysis. Interv Neuroradiol. 2021 Aug;27(4):577-583. doi: 10.1177/1591019921990962. Epub 2021 Feb 1. PMID 33525919
- [Background] Srivatsan A, Mohanty A, Nascimento FA, Hafeez MU, Srinivasan VM, Thomas A, Chen SR, Johnson JN, Kan P. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma: Meta-Analysis and Systematic Review. World Neurosurg. 2019 Feb;122:613-619. doi: 10.1016/j.wneu.2018.11.167. Epub 2018 Nov 24. PMID 30481628
- [Background] Sattari SA, Yang W, Shahbandi A, Feghali J, Lee RP, Xu R, Jackson C, Gonzalez LF, Tamargo RJ, Huang J, Caplan JM. Middle Meningeal Artery Embolization Versus Conventional Management for Patients With Chronic Subdural Hematoma: A Systematic Review and Meta-Analysis. Neurosurgery. 2023 Jun 1;92(6):1142-1154. doi: 10.1227/neu.0000000000002365. Epub 2023 Mar 17. PMID 36929762
- [Background] Ku JC, Dmytriw AA, Essibayi MA, Banihashemi MA, Vranic JE, Ghozy S, Altschul D, Regenhardt RW, Stapleton CJ, Yang VXD, Patel AB. Embolic Agent Choice in Middle Meningeal Artery Embolization as Primary or Adjunct Treatment for Chronic Subdural Hematoma: A Systematic Review and Meta-analysis. AJNR Am J Neuroradiol. 2023 Mar;44(3):297-302. doi: 10.3174/ajnr.A7796. Epub 2023 Feb 16. PMID 36797028
- [Background] Kan P, Maragkos GA, Srivatsan A, Srinivasan V, Johnson J, Burkhardt JK, Robinson TM, Salem MM, Chen S, Riina HA, Tanweer O, Levy EI, Spiotta AM, Kasab SA, Lena J, Gross BA, Cherian J, Cawley CM, Howard BM, Khalessi AA, Pandey AS, Ringer AJ, Hanel R, Ortiz RA, Langer D, Kelly CM, Jankowitz BT, Ogilvy CS, Moore JM, Levitt MR, Binning M, Grandhi R, Siddiq F, Thomas AJ. Middle Meningeal Artery Embolization for Chronic Subdural Hematoma: A Multi-Center Experience of 154 Consecutive Embolizations. Neurosurgery. 2021 Jan 13;88(2):268-277. doi: 10.1093/neuros/nyaa379. PMID 33026434
- [Background] Enriquez-Marulanda A, Gomez-Paz S, Salem MM, Mallick A, Motiei-Langroudi R, Arle JE, Stippler M, Papavassiliou E, Alterman RL, Ogilvy CS, Moore JM, Thomas AJ. Middle Meningeal Artery Embolization Versus Conventional Treatment of Chronic Subdural Hematomas. Neurosurgery. 2021 Aug 16;89(3):486-495. doi: 10.1093/neuros/nyab192. PMID 34171921
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660